CLINICAL TRIAL: NCT04327388
Title: An Adaptive Phase 3, Randomized, Double-blind, Placebo-controlled Study Assessing Efficacy and Safety of Sarilumab for Hospitalized Patients With COVID19
Brief Title: Sarilumab COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC16844; 2020-001162-12 (EudraCT Number); U1111-1249-6021 (Other: WHO Universal Trial Reference Number)
Record Dates: First submitted 2020-03-26; First posted 2020-03-31 (Actual); Results first posted 2021-05-13 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Corona Virus Infection
MeSH Terms: conditions — Coronavirus Infections | interventions — sarilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Sarilumab 200 mg (Experimental): Sarilumab 200 milligrams (mg), single dose of intravenous (IV) injection on Day 1. Participants could receive a second dose of sarilumab 200 mg 24 to 48 hours after the first dose if first and any one of last three criteria was met as compared to Day 1 (as per following protocol amendment 2 [dated 08-Apr-2020]):
  * Benefit risk assessment by the investigator favored the administration of another dose of study drug without compromising safety and
  * Increase/recurrence of fever or
  * Increase/no change in fraction of inspired oxygen (FiO2) requirement or
  * Required vasopressors, extracorporeal membrane oxygenation (ECMO) or development of multi-organ dysfunction.
  Interventions: Drug: Sarilumab SAR153191
- Sarilumab 400 mg (Experimental): Sarilumab 400 mg, single dose of IV injection on Day 1. Participants could receive a second dose of sarilumab 400 mg 24 to 48 hours after the first dose if first and any one of last three criteria was met as compared to Day 1 (as per following protocol amendment 2 [dated 08-Apr-2020]):
  * Benefit risk assessment by the investigator favored the administration of another dose of study drug without compromising safety and
  * Increase/recurrence of fever or
  * Increase/no change in FiO2 requirement or
  * Required vasopressors, ECMO or development of multi-organ dysfunction.
  Interventions: Drug: Sarilumab SAR153191
- Placebo (Placebo Comparator): Placebo (for sarilumab), single dose of IV injection on Day 1. Participants could receive a second dose of placebo (for sarilumab) 24 to 48 hours after the first dose if first and any one of last three criteria was met as compared to Day 1 (as per following protocol amendment 2 [dated 08-Apr-2020]):
  * Benefit risk assessment by the investigator favored the administration of another dose of study drug without compromising safety and
  * Increase/recurrence of fever or
  * Increase/no change in FiO2 requirement or
  * Required vasopressors, ECMO or development of multi-organ dysfunction.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sarilumab SAR153191 — Pharmaceutical form: Solution for injection Route of administration: Intravenous infusion
  Other Names: REGN88; Kevzara®
  Arms: Sarilumab 200 mg; Sarilumab 400 mg
Drug: Placebo — Pharmaceutical form: Solution for injection Route of administration: Intravenous infusion
  Arms: Placebo

SUMMARY:
Primary Objective:

To evaluate the clinical efficacy of sarilumab relative to the control arm in adult participants hospitalized with severe or critical Coronavirus Disease 2019 (COVID-19).

Secondary Objectives:

* Evaluate the 28-day survival rate.
* Evaluate the clinical efficacy of sarilumab compared to the control arm by clinical severity.
* Evaluate changes in the National Early Warning Score 2.
* Evaluate the duration of predefined symptoms and signs (if applicable).
* Evaluate the duration of supplemental oxygen dependency (if applicable).
* Evaluate the incidence of new mechanical ventilation use during the study.
* Evaluate the duration of new mechanical ventilation use during the Study.
* Evaluate the proportion of participants requiring rescue medication during the 28-day period.
* Evaluate need for admission into intensive care unit.
* Evaluate duration of hospitalization (days).
* The secondary safety objectives of the study were to evaluate the safety of sarilumab through hospitalization (up to Day 29 if participant was still hospitalized) compared to the control arm as assessed by incidence of:

  * Serious adverse events.
  * Major or opportunistic bacterial or fungal infections in participants with grade 4 neutropenia.
  * Grade greater than or equal to (>=) 2 infusion related reactions.
  * Grade >=2 hypersensitivity reactions.
  * Increase in alanine transaminase (ALT) >=3X upper limit of normal (ULN) (for participants with normal baseline) or greater than 3X ULN AND at least 2-fold increase from baseline value (for participants with abnormal baseline).
  * Major or opportunistic bacterial or fungal infections.

DETAILED DESCRIPTION:
An individual participant would complete the study approximately 60 days from screening to follow-up on day 60 ±7 days.

ELIGIBILITY:
Inclusion criteria :

Participants must be >=18 years of age. Participants must be hospitalized for less than or equal to 7 days with evidence of pneumonia and have one of the following disease categories: severe disease or critical disease.

Laboratory-confirmed severe acute respiratory syndrome coronavirus 2 infection.

Exclusion criteria:

Unlikely to survive after 48 hours from screening or unlikely to remain at the investigational site beyond 48 hours. Participants with multi organ dysfunction or requiring extracorporeal life support or renal replacement therapy were excluded.

Presence of neutropenia less than 2000/cubic millimeter (mmˆ3), aspartate transaminase or ALT greater than 5X ULN, platelets less than 50,000/mmˆ3.

Prior immunosuppressive therapies. Use of systemic chronic corticosteroids for non-COVID-19 related condition. Known or suspected history of tuberculosis. Suspected or known active systemic bacterial or fungal infections.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2020-03-28 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (47):
- Argentina (3):
  - Investigational Site Number 0320001, Caba
  - Investigational Site Number 0320003, Caba
  - Investigational Site Number 0320004, Caba
- Brazil (5):
  - Investigational Site Number 0760003, Porto Alegre
  - Investigational Site Number 0760004, São José do Rio Preto
  - Investigational Site Number 0760001, São Paulo
  - Investigational Site Number 0760002, São Paulo
  - Investigational Site Number 0760005, São Paulo
- Canada (5):
  - Investigational Site Number 1240001, Montreal
  - Investigational Site Number 1240005, Montreal
  - Investigational Site Number 1240004, Toronto
  - Investigational Site Number 1240002, Toronto
  - Investigational Site Number 1240003, Vancouver
- Chile (4):
  - Investigational Site Number 1520003, Santiago
  - Investigational Site Number 1520002, Santiago
  - Investigational Site Number 1520004, Santiago
  - Investigational Site Number 1520001, Talca
- France (7):
  - Investigational Site Number 2500001, Bordeaux
  - Investigational Site Number 2500007, Clamart
  - Investigational Site Number 2500006, La Roche-sur-Yon
  - Investigational Site Number 2500002, Nantes
  - Investigational Site Number 2500005, Paris
  - Investigational Site Number 2500003, Strasbourg
  - Investigational Site Number 2500004, Suresnes
- Germany (3):
  - Investigational Site Number 2760004, Cologne
  - Investigational Site Number 2760002, Essen
  - Investigational Site Number 2760001, Münster
- Israel (3):
  - Investigational site number 3760003, Ashdod
  - Investigational Site Number 3760002, Jerusalem
  - Investigational Site Number 3760001, Ramat Gan
- Italy (6):
  - Investigational Site Number 3800005, Milan
  - Investigational Site Number 3800001, Milan
  - Investigational Site Number 3800002, Milan
  - Investigational Site Number 3800003, Modena
  - Investigational Site Number 3800004, Parma
  - Investigational Site Number 3800006, Rozzano
- Japan (3):
  - Investigational Site Number 3920002, Fuchu-Shi
  - Investigational Site Number 3920003, Iruma-Gun
  - Investigational Site Number 3920001, Kamakura-Shi
- Russia (3):
  - Investigational Site Number 6430003, Moscow
  - Investigational Site Number 6430002, Moscow
  - Investigational Site Number 6430001, Moscow
- Spain (5):
  - Investigational Site Number 7240003, Barcelona
  - Investigational Site Number 7240004, Barcelona
  - Investigational Site Number 7240002, Madrid
  - Investigational Site Number 7240005, Madrid
  - Investigational Site Number 7240001, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Lescure FX, Honda H, Fowler RA, Lazar JS, Shi G, Wung P, Patel N, Hagino O; Sarilumab COVID-19 Global Study Group. Sarilumab in patients admitted to hospital with severe or critical COVID-19: a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Respir Med. 2021 May;9(5):522-532. doi: 10.1016/S2213-2600(21)00099-0. Epub 2021 Mar 4. PMID 33676590
- See also: EFC16844 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25257&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 46 active centers in 11 countries. A total of 431 participants were screened between 28 March 2020 and 02 July 2020, of which 10 participants were screen failures and 1 participant was randomized twice and thus excluded. Therefore, a total of 420 participants were randomized in the study treatment by the interactive response technology (IRT) (2:2:1 ratio) to receive sarilumab 200 milligrams (mg)/400 mg and placebo. Screen failures were mainly due to exclusion criteria met.
Pre-assignment Details: Randomization was stratified by severity of illness (severe disease, critical disease) and use of systemic corticosteroids (Yes/No).
Groups:
- Sarilumab 200 mg: Sarilumab 200 mg, single dose of intravenous (IV) injection on Day 1. Participants could receive a second dose of sarilumab 200 mg 24 to 48 hours after the first dose if first and any one of last three criteria was met as compared to Day 1 (as per following protocol amendment 2 [dated 08-Apr-2020]):
  * Benefit risk assessment by the investigator favored the administration of another dose of study drug without compromising safety and
  * Increase/recurrence of fever or
  * Increase/no change in fraction of inspired oxygen (FiO2) requirement or
  * Required vasopressors, extracorporeal membrane oxygenation (ECMO) or development of multi-organ dysfunction.
Period: Overall Study
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Started | 161 | 173 | 86
Treated | 159 | 173 | 84
Participants Who Received Second Dose (Participants who met prespecified criteria as per protocol amendment 2, received a second dose of the study drug (based on the original treatment group assigned) 24 to 48 hours after the first dose.) | 13 | 11 | 5
Completed | 141 | 153 | 75
Not Completed | 20 | 20 | 11
Not completed — Adverse Event | 17 | 18 | 9
Not completed — Other | 1 | 2 | 0
Not completed — Randomized and not treated | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized population.
Groups:
- Sarilumab 200 mg: Sarilumab 200 mg, single dose of IV injection on Day 1. Participants could receive a second dose of sarilumab 200 mg 24 to 48 hours after the first dose if first and any one of last three criteria was met as compared to Day 1 (as per following protocol amendment 2 [dated 08-Apr-2020]):
  * Benefit risk assessment by the investigator favored the administration of another dose of study drug without compromising safety and
  * Increase/recurrence of fever or
  * Increase/no change in FiO2 requirement or
  * Required vasopressors, ECMO or development of multi-organ dysfunction.
- Total: Total of all reporting groups
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo | Total
Number analyzed (Participants) | 161 | 173 | 86 | 420
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (13.7) | 58.0 (14.1) | 59.9 (14.8) | 58.5 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 74 | 30 | 156
  Male | 109 | 99 | 56 | 264
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 1 | 5
  Asian | 5 | 9 | 6 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 3 | 5 | 1 | 9
  White | 128 | 128 | 69 | 325
  More than one race | 0 | 3 | 0 | 3
  Unknown or Not Reported | 23 | 26 | 8 | 57
Clinical Status: 7-point ordinal scale [Count of Participants; unit: Participants] — 7-point ordinal scale with scores range from: 1= death; 2= hospitalized, on invasive mechanical ventilation/ECMO; 3= hospitalized, on non-invasive ventilation/high flow oxygen devices; 4= hospitalized, requiring supplemental oxygen; 5= hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (Coronavirus Disease 2019 [COVID-19] related/otherwise); 6= hospitalized, not requiring supplemental oxygen - no longer required ongoing medical care; 7= not hospitalized, higher score = less severity. Number of participants in each scale category were reported.
  Participants
    Scale Score 1 | 0 | 0 | 0 | 0
    Scale Score 2 | 17 | 24 | 10 | 51
    Scale Score 3 | 28 | 21 | 11 | 60
    Scale Score 4 | 113 | 128 | 65 | 306
    Scale Score 5 | 3 | 0 | 0 | 3
    Scale Score 6 | 0 | 0 | 0 | 0
    Scale Score 7 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Improvement in Clinical Status of Participants (Using 7-point Ordinal Scale Score) by at Least 2 Points
Description: Time to improvement of greater than or equal (>=) 2 points in clinical status assessment was defined as time (in days) from first dose of study drug to the time of first occurrence of improvement of >=2 points in clinical status of participants assessed using 7-point ordinal scale (calculated as: Date of first occurrence/episode of the event - date of first dose + 1). Seven-point ordinal scale for clinical assessment ranges from 1= death; 2= hospitalized, on invasive mechanical ventilation/ECMO; 3= hospitalized, on non-invasive ventilation/high flow oxygen devices; 4= hospitalized, requiring supplemental oxygen; 5= hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related/otherwise); 6= hospitalized, not requiring supplemental oxygen - no longer required ongoing medical care; 7= not hospitalized, higher score = less severity. Kaplan-Meier method was used for analysis.
Time Frame: Baseline to Day 29
Population: Analysis was performed on modified intention-to-treat (mITT) population which included all participants who were treated with study medication and were analyzed according to the initial treatment assigned to the participant (as randomized).
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 159 | 173 | 84
days | 10.0 [9.00 to 12.00] | 10.0 [9.00 to 13.00] | 12.0 [9.00 to 15.00]
Statistical Analysis 1: Comparison: Sarilumab 200 mg vs Placebo; Test type: Superiority; p = 0.9561, Log-rank test; Analyzed based on logrank test stratified by severity of illness (severe, critical) and use of systemic corticosteroids (Yes, No) as entered in IRT; Hazard Ratio (HR) = 1.026, 95% CI 2-sided [0.751 to 1.402] — Hazard ratio for estimation of treatment effect of each sarilumab dose versus placebo was assessed by cox proportional hazard model stratified by severity of illness (severe, critical) and use of systemic corticosteroids (Yes, No) as entered in IRT
Statistical Analysis 2: Comparison: Sarilumab 400 mg vs Placebo; Test type: Superiority; p = 0.3376, Log-rank test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.135, 95% CI 2-sided [0.835 to 1.543] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Percentage of Participants Who Were Alive at Day 29
Description: Percentage of participants who were alive at Day 29 were reported in this outcome measure.
Time Frame: Day 29
Population: Analysis was performed on mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 159 | 173 | 84
percentage of participants | 89.9 | 91.9 | 91.7
Statistical Analysis 1: Comparison: Sarilumab 200 mg vs Placebo; Test type: Superiority; p = 0.6280, Cochran-Mantel-Haenszel; By Cochran-Mantel-Haenszel test stratified by severity of illness (severe, critical) and use of systemic corticosteroids (Yes, No) as entered in IRT; Difference in percentage = -1.7, 95% CI 2-sided [-9.27 to 5.81]
Statistical Analysis 2: Comparison: Sarilumab 400 mg vs Placebo; Test type: Superiority; p = 0.8478, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Difference in percentage = 0.2, 95% CI 2-sided [-6.93 to 7.41]

3. Secondary Outcome: Percentage of Participants With Improvement in Clinical Status (According to 7-point Ordinal Scale Score) by at Least 1 Point From Baseline at Days 4, 7, 15, 21, and 29
Description: Clinical status of participants was assessed using 7-point ordinal scale ranges from: 1= death; 2= hospitalized, on invasive mechanical ventilation/ECMO; 3= hospitalized, on non-invasive ventilation/high flow oxygen devices; 4= hospitalized, requiring supplemental oxygen; 5= hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related/otherwise); 6= hospitalized, not requiring supplemental oxygen - no longer required ongoing medical care; 7= not hospitalized, higher score=less severity. Percentage of participants With >=1 point improvement in clinical status from Baseline at Days 4, 7, 15, 21, and 29 (assessed using the 7-point ordinal scale) were reported.
Time Frame: Baseline, Days 4, 7, 15, 21, and 29
Population: Analysis was performed on mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 159 | 173 | 84
percentage of participants
  Day 4 | 25.2 | 25.4 | 23.8
  Day 7 | 51.6 | 48.6 | 42.9
  Day 15 | 74.8 | 76.9 | 71.4
  Day 21 | 80.5 | 81.5 | 85.7
  Day 29 | 84.9 | 84.4 | 88.1

4. Secondary Outcome: Change From Baseline at Days 4, 7, 15, 21, 29 in 7-point Ordinal Scale Score
Description: Clinical status of participants was assessed using 7-point ordinal scale ranges from: 1= death; 2= hospitalized, on invasive mechanical ventilation/ECMO; 3= hospitalized, on non-invasive ventilation/high flow oxygen devices; 4= hospitalized, requiring supplemental oxygen; 5= hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related/otherwise); 6= hospitalized, not requiring supplemental oxygen - no longer required ongoing medical care; 7= not hospitalized, higher score=less severity.
Time Frame: Baseline, Days 4, 7, 15, 21, and 29
Population: Analysis was performed on mITT population. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 159 | 173 | 84
scores on a scale
  Day 4 | 0.1 (0.9) | 0.1 (1.0) | 0.2 (0.9)
  Day 7 | 0.7 (1.5) | 0.7 (1.6) | 0.7 (1.4)
  Day 15: number analyzed (Participants) | 158 | 171 | 83
  Day 15 | 1.9 (1.8) | 2.0 (1.9) | 1.7 (1.8)
  Day 21: number analyzed (Participants) | 155 | 169 | 83
  Day 21 | 2.3 (1.9) | 2.3 (1.9) | 2.5 (1.7)
  Day 29: number analyzed (Participants) | 156 | 170 | 83
  Day 29 | 2.5 (1.9) | 2.5 (1.9) | 2.7 (1.6)

5. Secondary Outcome: Time to Resolution of Fever
Description: Resolution of fever was defined as body temperature less than or equal to (<=) 36.6 degree Celsius (°C) (axilla), or <=37.2°C (oral), or <=37.8°C (rectal or tympanic) for at least 48 hours without antipyretics/until discharge, whichever was sooner. Time to resolution of fever (in days) was calculated as: date of first occurrence/episode of the event (resolution of fever) - date of first dose + 1. Kaplan-Meier method was used for estimation.
Time Frame: Baseline to Day 29
Population: Analysis was performed on mITT population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 159 | 173 | 84
days | 8.0 [7.00 to 9.00] | 9.0 [7.00 to 10.00] | 7.0 [6.00 to 12.00]

6. Secondary Outcome: Time to Resolution of Fever and Improvement in Oxygenation
Description: Time to resolution of fever was defined as body temperature <=36.6°C (axilla), or <=37.2 °C (oral), or <=37.8°C (rectal or tympanic) for at least 48 hours without antipyretics or until discharge, whichever was sooner. Improvement in oxygenation was defined as oxygen saturation (SpO2)/FiO2 of 50 or greater compared to the nadir SpO2/FiO2 for at least 48 hours, or until discharge, whichever was sooner. Nadir SpO2/FiO2 was the nadir (lowest value) at any point in the study. Time to resolution of fever and improvement in oxygenation (in days) was calculated as: date of first occurrence/episode of the event (resolution of fever and improvement in oxygenation) - date of first dose + 1. Kaplan-Meier method was used for estimation.
Time Frame: Baseline to Day 29
Population: Analysis was performed on mITT population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 159 | 173 | 84
days | 9.0 [8.00 to 10.00] | 10.0 [9.00 to 13.00] | 8.0 [7.00 to 12.00]

7. Secondary Outcome: Number of Days With Fever
Description: Fever was defined as body temperature greater than (>) 37.4°C (axilla), or >38.0 °C (oral), or >38.4°C (rectal or tympanic) based on maximum value observed during a 24-hour period. Number of days with fever were reported. Least square (LS) mean and standard error (SE) were estimated using the analysis of covariance (ANCOVA) model with treatment group and randomization strata as fixed effects.
Time Frame: Baseline to Day 29
Population: Analysis was performed on mITT population. Here, overall number of participants analyzed = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 143 | 159 | 77
days | 1.2 (0.23) | 1.3 (0.21) | 1.8 (0.30)

8. Secondary Outcome: Percentage of Participants in Each National Early Warning Score 2 (NEWS2) Clinical Risk Category at Baseline and at Days 4, 7, 15, 21, and 29
Description: NEWS2: used to standardize assessment of acute-illness severity, track clinical condition of participants and to alert clinical teams to participant deterioration. NEWS2 score was based on 7 clinical parameters: respiration rate, oxygen saturation, supplemental oxygen, systolic blood pressure, pulse rate, level of consciousness, and temperature. A score of 0, 1, 2, and 3 was allocated to each parameter except supplemental oxygen (a score of 0 or 1 was allocated) and level of consciousness (a score of 0 or 3 was allocated), where 0 = normal health condition to 3 = worst health condition; higher score indicated more severity. All scores were summed to get an aggregate score. Aggregate NEWS2 score ranged from 0 to 19, with higher scores meaning more severity/higher risk. Percentage of participants in following clinical risk categories were reported: low risk (score 0 to 4); low to medium risk (score of 3 in any individual parameter); medium risk (score 5 to 6); high risk (score 7 to 19).
Time Frame: Baseline, Days 4, 7, 15, 21, and 29
Population: Analysis was performed on mITT population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Number; unit: percentage of participants
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 159 | 169 | 84
percentage of participants
  Baseline: Low: number analyzed (Participants) | 146 | 163 | 79
  Baseline: Low | 28.8 | 22.1 | 34.2
  Baseline: Low to Medium: number analyzed (Participants) | 146 | 163 | 79
  Baseline: Low to Medium | 0 | 0 | 0
  Baseline: Medium: number analyzed (Participants) | 146 | 163 | 79
  Baseline: Medium | 34.2 | 37.4 | 27.8
  Baseline: High: number analyzed (Participants) | 146 | 163 | 79
  Baseline: High | 37.0 | 40.5 | 38.0
  Day 4: Low | 52.8 | 56.2 | 40.5
  Day 4: Low to Medium | 0.6 | 1.2 | 0
  Day 4: Medium | 19.5 | 16.6 | 28.6
  Day 4: High | 27.0 | 26.0 | 31.0
  Day 7: Low: number analyzed (Participants) | 135 | 143 | 74
  Day 7: Low | 57.0 | 60.8 | 51.4
  Day 7: Low to Medium: number analyzed (Participants) | 135 | 143 | 74
  Day 7: Low to Medium | 0 | 2.1 | 0
  Day 7: Medium: number analyzed (Participants) | 135 | 143 | 74
  Day 7: Medium | 20.0 | 10.5 | 20.3
  Day 7: High: number analyzed (Participants) | 135 | 143 | 74
  Day 7: High | 23.0 | 26.6 | 28.4
  Day 15: Low: number analyzed (Participants) | 61 | 67 | 36
  Day 15: Low | 52.5 | 52.2 | 61.1
  Day 15: Low to Medium: number analyzed (Participants) | 61 | 67 | 36
  Day 15: Low to Medium | 0 | 1.5 | 2.8
  Day 15: Medium: number analyzed (Participants) | 61 | 67 | 36
  Day 15: Medium | 21.3 | 19.4 | 13.9
  Day 15: High: number analyzed (Participants) | 61 | 67 | 36
  Day 15: High | 26.2 | 26.9 | 22.2
  Day 21: Low: number analyzed (Participants) | 29 | 38 | 12
  Day 21: Low | 44.8 | 50.0 | 66.7
  Day 21: Low to Medium: number analyzed (Participants) | 29 | 38 | 12
  Day 21: Low to Medium | 13.8 | 0 | 0
  Day 21: Medium: number analyzed (Participants) | 29 | 38 | 12
  Day 21: Medium | 24.1 | 21.1 | 8.3
  Day 21: High: number analyzed (Participants) | 29 | 38 | 12
  Day 21: High | 17.2 | 28.9 | 25.0
  Day 29: Low: number analyzed (Participants) | 14 | 18 | 5
  Day 29: Low | 57.1 | 27.8 | 60.0
  Day 29: Low to Medium: number analyzed (Participants) | 14 | 18 | 5
  Day 29: Low to Medium | 0 | 0 | 0
  Day 29: Medium: number analyzed (Participants) | 14 | 18 | 5
  Day 29: Medium | 14.3 | 27.8 | 20.0
  Day 29: High: number analyzed (Participants) | 14 | 18 | 5
  Day 29: High | 28.6 | 44.4 | 20.0

9. Secondary Outcome: Time to National Early Warning Score of Less Than (<) 2 and Maintained for 24 Hours
Description: Time to NEWS2 <2 and maintained for 24 hours: time (in days) from 1st dose of study drug until 1st occurrence of NEWS score of <2 (maintained for 24 hours); calculated as: date of 1st occurrence/episode of event (NEWS score of <2) - date of 1st dose + 1. NEWS2 score was based on 7 clinical parameters: respiration rate, oxygen saturation, supplemental oxygen, systolic blood pressure, pulse rate, level of consciousness, and temperature. A score of 0, 1, 2, and 3 was allocated to each parameter except supplemental oxygen (score of 0 or 1 was allocated) and level of consciousness (score of 0 or 3 was allocated), where 0=normal health condition to 3=worst health condition; higher score=more severity. All scores were summed to get an aggregate score which ranged from 0 to 19, with higher scores=more severity/higher risk. Kaplan-Meier method was used for analysis.
Time Frame: Baseline to Day 29
Population: Analysis was performed on mITT population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 159 | 173 | 84
days | 9.0 [7.00 to 10.00] | 9.0 [8.00 to 11.00] | 11.0 [8.00 to 14.00]

10. Secondary Outcome: Change From Baseline at Days 4, 7, 15, 21, and 29 in National Early Warning Score 2
Description: The NEWS2 was used to standardize the assessment of acute-illness severity, track the clinical condition of participants, and to alert clinical teams to participant deterioration. NEWS2 score is based on 7 clinical parameters: respiration rate, oxygen saturation, supplemental oxygen, systolic blood pressure, pulse rate, level of consciousness, and temperature. A score of 0, 1, 2, and 3 was allocated to each parameter except supplemental oxygen (a score of 0 or 1 was allocated) and level of consciousness (a score of 0 or 3 was allocated), where 0 = normal health condition to 3 = worst health condition; higher score indicated more severity. All scores were summed to get an aggregate score. Aggregate NEWS2 score ranged from 0 to 19, with higher scores meaning more severity/higher risk. LS means and SE were estimated using ANCOVA model with treatment group and randomization strata as fixed effects, and baseline NEWS2 score as a covariate.
Time Frame: Baseline, Days 4, 7, 15, 21, and 29
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 146 | 159 | 79
scores on a scale
  Day 4 | -1.07 (0.212) | -1.25 (0.198) | -0.36 (0.274)
  Day 7: number analyzed (Participants) | 122 | 133 | 69
  Day 7 | -1.63 (0.265) | -1.47 (0.245) | -0.83 (0.338)
  Day 15: number analyzed (Participants) | 55 | 62 | 33
  Day 15 | -2.10 (0.508) | -1.83 (0.467) | -2.36 (0.641)
  Day 21: number analyzed (Participants) | 26 | 34 | 12
  Day 21 | -3.02 (0.769) | -2.24 (0.676) | -2.96 (1.090)
  Day 29: number analyzed (Participants) | 13 | 17 | 5
  Day 29 | -2.57 (0.936) | -1.27 (0.884) | -3.64 (1.508)

11. Secondary Outcome: Time-to-improvement in Oxygenation
Description: Time-to-improvement in oxygenation was defined as increase in SpO2/FiO2 of 50 or greater compared to the nadir SpO2/FiO2 for at least 48 hours or until discharge, whichever was sooner. Nadir SpO2/FiO2 was the nadir (lowest value) at any point in the study. Time to improvement in oxygenation was calculated as: date of first occurrence/episode of the event (oxygenation) - date of first dose + 1. Kaplan-Meier method was used for estimation.
Time Frame: Baseline to Day 29
Population: Analysis was performed on mITT population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 159 | 173 | 84
days | 6.0 [5.00 to 7.00] | 6.0 [5.00 to 7.00] | 7.0 [5.00 to 8.00]

12. Secondary Outcome: Percentage of Participants Alive Off Supplemental Oxygen at Day 29
Description: Supplemental oxygen was defined as oxygen administration by nasal cannula, simple face mask, or other similar oxygen delivery device.
Time Frame: Day 29
Population: Analysis was performed on mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 159 | 173 | 84
percentage of participants | 84.9 | 83.8 | 86.9

13. Secondary Outcome: Percentage of Days With Hypoxemia
Description: Hypoxemia (low level of oxygen in the blood) was defined as SpO2 <93% on room air, or required supplemental oxygen, or mechanical ventilatory support. Days meeting the criteria for hypoxemia since the first study dose were counted and the percentage of days with hypoxemia were calculated as:100*number of days with the hypoxemia divided by number of days of follow up (defined as the earlier date of death or discharge or last visit up to Day 29). LS mean and SE were estimated using the ANCOVA model with treatment group and randomization strata as fixed effects.
Time Frame: Baseline to Day 29
Population: Analysis was performed on mITT population.
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 159 | 173 | 84
percentage of days | 73.01 (2.063) | 75.10 (1.941) | 76.32 (2.724)

14. Secondary Outcome: Percentage of Days With Supplemental Oxygen Use
Description: Supplemental oxygen (oxygen therapy) was defined as oxygen administration using oxygen delivery device (e.g. nasal cannula, simple face mask, non-rebreather mask, high flow nasal cannula, non-invasive ventilation, invasive mechanical ventilation, extracorporeal life support, etc.). Days meeting the criteria for supplemental oxygen use since the first study dose were counted and the percentage of days with supplemental oxygen use were calculated as:100*number of days with the supplemental oxygen use divided by number of days of follow up (defined as the earlier date of death or discharge or last visit up to Day 29) . LS mean and SE were estimated using the ANCOVA model with treatment group and randomization strata as fixed effects.
Time Frame: Baseline to Day 29
Population: Analysis was performed on mITT population.
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 159 | 173 | 84
percentage of days | 70.57 (2.082) | 73.30 (1.959) | 73.23 (2.748)

15. Secondary Outcome: Percentage of Days With Resting Respiratory Rate > 24 Breaths Per Minute
Description: Resting respiratory rate was measured in terms of number of breaths per minute (bpm) while a person is at rest. Only the days with respiratory rate >24 breath per minute since the first dose were counted and percentage of days with respiratory rate > 24 bpm were calculated as:100*number of days with respiratory rate >24 bpm divided by number of days of follow up (defined as the earlier date of death or discharge or last visit up to Day 29). LS mean and SE were estimated using the ANCOVA model with treatment group and randomization strata as fixed effects.
Time Frame: Baseline to Day 29
Population: Analysis was performed on mITT population. Hence, overall number of participants analyzed = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 150 | 164 | 78
percentage of days | 14.74 (1.582) | 14.58 (1.485) | 15.74 (2.105)

16. Secondary Outcome: Time to Oxygen Saturation >= 94% on Room Air
Description: Time to oxygen saturation >=94% on room air was defined as the time (in days) from first dose of study drug until the time of first occurrence of oxygen saturation >=94% and it was calculated as: Date of first occurrence/episode of the event (oxygen saturation >=94%) - date of first dose + 1.Kaplan-Meier method was used for estimation.
Time Frame: Baseline to Day 29
Population: Analysis was performed on mITT population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 159 | 173 | 84
days | 8.0 [6.00 to 10.00] | 8.0 [8.00 to 11.00] | 8.0 [7.00 to 11.00]

17. Secondary Outcome: Mean Number of Ventilator Free Days
Description: Mean number of ventilator free days in participants were reported.
Time Frame: Baseline to Day 29
Population: Analysis was performed on mITT population.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 159 | 173 | 84
days | 23.8 (9.4) | 24.0 (8.8) | 24.9 (8.6)

18. Secondary Outcome: Percentage of Participants With Initiation of Mechanical Ventilation, Non-invasive Ventilation, or Use of High Flow Nasal Cannula
Description: Percentage of participants With initiation of mechanical ventilation or non-invasive ventilation, or use of high flow nasal cannula were reported in this outcome measure.
Time Frame: Baseline to Day 29
Population: Analysis was performed on mITT population. Here, "overall number of participants analyzed" = participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 127 | 141 | 68
percentage of participants | 20.5 | 23.4 | 19.1

19. Secondary Outcome: Percentage of Participants Who Required Rescue Medication
Description: Rescue medications were defined as the immunosuppressive (methylprednisolone, dexamethasone and prednisone) therapies. During the course of the study, participant who required rescue therapy was based on the judgement of the study physician.
Time Frame: Baseline to Day 28
Population: Analysis was performed on mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 159 | 173 | 84
percentage of participants | 13.8 | 15.0 | 22.6

20. Secondary Outcome: Percentage of Participants Who Needed Intensive Care Unit (ICU) Care During Study
Description: Percentage of participants who needed ICU care until Day 29 were reported for those not in an ICU at baseline.
Time Frame: Baseline to Day 29
Population: Analysis was performed on mITT population. Here, "overall number of participants analyzed"=participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 98 | 114 | 56
percentage of participants | 11.2 | 14.9 | 12.5

21. Secondary Outcome: Number of Days of Hospitalization Among Survivors (Alive Participants)
Description: Number of days of hospitalization among alive participants were counted at Day 60 since the first dose. LS mean and SE were estimated using the ANCOVA model with treatment group and randomization strata as fixed effects.
Time Frame: At Day 60
Population: as for outcome 20
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 142 | 155 | 75
days | 15.6 (0.96) | 16.1 (0.91) | 15.9 (1.27)

22. Secondary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (SAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily had to have a causal relationship with the treatment. Treatment-emergent AEs (TEAEs) were the AEs that developed or worsened or became serious during the TEAE period (from the time of first dose of study drug to the last dose of study drug + 60 days). SAEs were any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event.
Time Frame: Baseline up to 60 days
Population: Analysis was performed on safety population which included all randomized participants who were treated with the study medication and were analyzed according to the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 159 | 173 | 84
Participants | 42 | 51 | 20

23. Secondary Outcome: Number of Participants With Major or Opportunistic Bacterial or Fungal Infections
Description: Major or opportunistic bacterial or fungal infections was considered as an adverse event of special interest (AESI: defined as an AE [serious or non-serious] of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the Investigator to the Sponsor was required).
Time Frame: Baseline up to 60 days
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 159 | 173 | 84
Participants | 8 | 15 | 3

24. Secondary Outcome: Number of Participants With Grade 4 Neutropenia and Grade 4 Neutropenia With Concurrent Invasive Infection
Description: Grade 4 neutropenia was defined as participants with absolute neutrophil count (ANC) <500 per cubic millimeter (mm^3). Grade 4 neutropenia with concurrent invasive infection was defined as infections and infestations (in participants with Grade 4 neutropenia) within 1 week of ANC <500/mm^3 and was considered as an AESI (defined as an AE [serious or non-serious] of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the Investigator to the Sponsor was required).
Time Frame: Baseline up to 60 days
Population: Analysis was performed on safety population. Here, 'number analyzed' = participants with available data for each specified category and "0" in the number analyzed field signifies that no participants had Grade 4 neutropenia and therefore were not evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 159 | 173 | 84
Participants
  Grade 4 neutropenia | 3 | 6 | 0
  Grade 4 neutropenia with concurrent invasive infection: number analyzed (Participants) | 3 | 6 | 0
  Grade 4 neutropenia with concurrent invasive infection | 0 | 0 |

25. Secondary Outcome: Number of Participants With Grade >=2 Infusion Reactions, Grade >=2 Hypersensitivity Reactions and Gastrointestinal Perforation
Description: Grade >=2 (moderate) infusion related reactions (defined as any TEAE signs or symptoms experienced by participants who received study medication within 24 hours of the start of infusion) and Grade >=2 (moderate) hypersensitivity reactions (anaphylactic reaction, hypersensitivity or angioedema and moderate reactions) were considered as AESI which was defined as an AE (serious or non-serious) of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the Investigator to the Sponsor was required. Gastrointestinal Perforation was defined as formation of a hole through the stomach, large bowel or small intestine.
Time Frame: Baseline up to 60 days
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 159 | 173 | 84
Participants
  Grade >=2 Infusion related reactions | 1 | 6 | 0
  Grade >=2 Hypersensitivity reactions | 1 | 7 | 0
  Gastrointestinal perforation | 1 | 0 | 0

26. Secondary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities (PCSA): Hematological Parameter - Hemoglobin, Leukocytes and Platelets
Description: Criteria for PCSA:
  * Hemoglobin: less than or equal to (<=) 115 grams per liter (g/L) (male) and <=95 g/L (female); greater than or equal to (>=) 185 g/L (male) and >=165 g/L (female); and decrease from baseline >=20 g/L.
  * Leukocytes: <3.0*10^9/Liters (L) (Non-Black) or <2.0*10^9/L (black); >=16.0*10^9/L.
  * Platelets: < 100*10^9/L; >=700*10^9/L.
Time Frame: Baseline up to 60 days
Population: Analysis was performed on safety population. Here, overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 156 | 170 | 84
Participants
  Hemoglobin <=115 g/L (male) and <=95 g/L (female) | 29 | 34 | 15
  Hemoglobin >=185 g/L (male) and >=165 g/L (female) | 0 | 0 | 0
  Hemoglobin decrease from baseline >=20 g/L | 32 | 30 | 15
  Leukocytes <3.0*10^9/L (Non-Black) or <2.0*10^9/L (black) | 19 | 31 | 1
  Leukocytes >=16*10^9/L | 13 | 21 | 6
  Platelets <100*10^9/L | 2 | 7 | 3
  Platelets >=700*10^9/L | 3 | 2 | 2

27. Secondary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Renal Function Parameters
Description: Criteria for PCSA: Creatinine: >=150 micromoles per liter (mcmol/L); >=30% change from baseline; >= 100% change from baseline.
Time Frame: Baseline up to 60 days
Population: as for outcome 26
Measure: Count of Participants; unit: Participants
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 156 | 170 | 84
Participants
  Creatinine >=150 mcmol/L | 15 | 15 | 5
  >=30% change from baseline in Creatinine | 31 | 30 | 10
  >=100% change from baseline in Creatinine | 6 | 7 | 3

28. Secondary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Liver Function Parameters
Description: * Alanine Aminotransferase (ALT): >3 upper limit of normal (ULN); >5 ULN; >10 ULN and >20 ULN.
  * Bilirubin: >1.5 ULN; >2 ULN.
Time Frame: Baseline up to 60 days
Population: Analysis was performed on safety population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
Number analyzed (Participants) | 156 | 169 | 84
Participants
  ALT >3 ULN: number analyzed (Participants) | 156 | 168 | 83
  ALT >3 ULN | 60 | 63 | 24
  ALT >5 ULN: number analyzed (Participants) | 156 | 168 | 83
  ALT >5 ULN | 28 | 25 | 12
  ALT >10 ULN: number analyzed (Participants) | 156 | 168 | 83
  ALT >10 ULN | 6 | 5 | 3
  ALT >20 ULN: number analyzed (Participants) | 156 | 168 | 83
  ALT >20 ULN | 1 | 0 | 0
  Bilirubin >1.5 ULN | 5 | 4 | 4
  Bilirubin >2 ULN | 4 | 2 | 2

ADVERSE EVENTS:
Time Frame: All AEs were collected from the time of first dose of study drug up to 60 days regardless of seriousness or relationship to study drug.
Description: Reported AEs and deaths were TEAEs that developed/worsened in grade or became serious during 'treatment-emergent adverse event period' (from the time of first dose of study drug to the last dose of study drug + 60 days). Analysis was performed on safety population.
Arm/Group | Sarilumab 200 mg | Sarilumab 400 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 17/159 | 18/173 | 9/84
Serious Adverse Events (participants affected / at risk) | 42/159 | 51/173 | 20/84
Other Adverse Events (participants affected / at risk) | 57/159 | 68/173 | 14/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sarilumab 200 mg (N=159) | Sarilumab 400 mg (N=173) | Placebo (N=84)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Blood Loss Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Intracardiac Thrombus (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pulseless Electrical Activity (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Entropion (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric Ulcer Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intra-Abdominal Haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Megacolon (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Multiple Organ Dysfunction Syndrome (General disorders) | 2 (2) | 3 (3) | 3 (3)
Physical Deconditioning (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic Steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Hepatitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatocellular Injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess Limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacterial Infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Covid-19 Pneumonia (Infections and infestations) | 11 (11) | 4 (4) | 2 (2)
Clostridium Difficile Colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis Klebsiella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower Respiratory Tract Infection Fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 6 (6) | 0 (0)
Pneumonia Bacterial (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Pneumonia Klebsiella (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic Shock (Infections and infestations) | 4 (4) | 4 (5) | 2 (2)
Soft Tissue Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Systemic Bacterial Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Systemic Candida (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 4 (4) | 3 (3) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Brain Oedema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Carotid Artery Thrombosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxic-Ischaemic Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2) | 4 (4) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Renal Impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Organising Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax Spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5) | 3 (3)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral Artery Occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis Superficial (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vena Cava Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Venous Thrombosis Limb (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sarilumab 200 mg (N=159) | Sarilumab 400 mg (N=173) | Placebo (N=84)
Neutropenia (Blood and lymphatic system disorders) | 11 (11) | 13 (13) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 48 (48) | 58 (59) | 14 (14)
Aspartate Aminotransferase Increased (Investigations) | 11 (11) | 15 (16) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/88/NCT04327388/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/88/NCT04327388/SAP_001.pdf